CLINICAL TRIAL: NCT02155608
Title: Developmental Pilot Study of External Trigeminal Nerve Stimulation for ADHD
Brief Title: Trigeminal Nerve Stimulation for ADHD
Acronym: TNS for ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James McGough, Professor of Clinical Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIMH R34MH101282; R34MH101282 (NIH)
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; neuromodulation; trigeminal nerve stimulation; cognition
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, sham-controlled.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active eTNS (Experimental): Following screening and determination of eligibility, participants at baseline are randomized to receive 4 weeks nightly treatment with active or sham eTNS, followed by one week ongoing blinded assessment following treatment discontinuation. Positive responders will be invited to participate in a 12-month open extension.
  Interventions: Device: Active eTNS
- Sham eTNS (Sham Comparator): Following screening and determination of eligibility, participants at baseline are randomized to receive 4 weeks nightly treatment with active or sham eTNS, followed by one week ongoing blinded assessment following treatment discontinuation. Following double-blind phase, interested participants randomized to sham have an option for a 4-week open TNS trial. Positive responders will be invited to participate in a 12-month open extension.
  Interventions: Device: Sham eTNS

INTERVENTIONS:
Device: Active eTNS — Participants will receive active trigeminal nerve stimulation (TNS) administered by the Monarch eTNS System nightly during sleep for 4 weeks, followed by one week of observation and followup while remaining blinded following treatment discontinuation. Participant deemed to be positive responders to blinded active treatment will be invited to continue open eTNS in a 12 month extension period.
  Other Names: Trigeminal Nerve Stimulation; Monarch eTNS SystemTM (NeuroSigma, Inc., Los Angeles CA
  Arms: Active eTNS
Device: Sham eTNS — Participants will receive sham trigeminal nerve stimulation (TNS) administered by the Monarch eTNS System nightly during sleep for 4 weeks, followed by one week of observation and followup while remaining blinded following treatment discontinuation. At the conclusion of the blinded trial, participants randomized to the sham group will be offered 4 weeks of open eTNS treatment. Participants deemed to be positive responders to open treatment will be invited to continue open nightly eTNS in a 12 month extension period.
  Arms: Sham eTNS

SUMMARY:
The purpose of this study is to develop external Trigeminal Nerve Stimulation (eTNS) as a potential nonmedication treatment for attention-deficit/hyperactivity disorder (ADHD).

Study hypothesis address potential differences over 4 weeks of active vs. sham eTNS treatment on ADHD symptoms, measures of executive function, electroencephalography (EEG) profiles, other dimensional measures of height, weight, mood, anxiety, and sleep, and side effect profiles.

DETAILED DESCRIPTION:
This three-year developmental study is a double-blind randomized trial of active vs. inactive sham eTNS for ADHD, with four weeks acute treatment followed by an additional one week of clinical observation and testing after treatment cessation.

The study will enroll 85-90 participants aged 8-12 years to achieve a completion target of N=36 for each study condition (total final N = 72). Participants will meet Diagnostic and Statistical Manual-5 (DSM-5) criteria for ADHD, any current presentation, as established by the Behavior Disorders Module of the Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS-PL) and clinical interview.

Other screening procedures include measures of ADHD symptom severity, other behavioral ratings, and cognitive assessments. Once inclusion/exclusion criteria have been reviewed and verified, participants in Phase 1A will have a pre-treatment visit to establish behavioral and cognitive baseline ratings and to obtain an EEG. Participants and parents will be instructed in the use of eTNS, and participants will begin use of the eTNS as directed during sleep each night. Participants will be randomized 1:1 to active or inactive sham eTNS. Participants, families, and most of the study team will remain blind to treatment assignment. Participants will have weekly assessments over the five-week study to assess behavioral, cognitive, and brain activation change and to monitor safety, tolerability, and compliance. Weekly ratings will be obtained from a parent, teacher, and clinician investigator. EEG will occur at baseline, end of treatment (week 4).

In Phase 1B, all participants remain blinded for one week after cessation of the intervention and return for a final visit to assess residual effects of eTNS therapy vs. sham.

ELIGIBILITY:
Inclusion Criteria:

* male and female children ages 8 to 12 years with DSM-5 ADHD, any current presentation, as determined by KSADS and clinical interview
* minimum scores of 12 on both the inattentive and hyperactive/impulsive subscales of the baseline ADHD-RS
* CGI-S score at baseline ≥ 4
* no current medication with CNS effects
* parents able and willing to monitor proper use of the stimulation device and complete all required rating scales
* estimated Full Scale IQ ≥ 85 based on WASI subtests
* parent and participant able to complete rating scales and other measures in English
* able to cooperate during EEG

Exclusion Criteria:

* impaired functioning to a degree that requires immediate initiation of ADHD medication in the opinion of the parents and/or investigator
* current diagnosis of autism spectrum disorder or major depression
* history of lifetime psychosis, mania, seizure disorder or head injury with loss of consciousness
* baseline suicidality

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J McGough, M.D., Principal Investigator — University of California, Los Angeles; Sandra K Loo, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McGough JJ, Sturm A, Cowen J, Tung K, Salgari GC, Leuchter AF, Cook IA, Sugar CA, Loo SK. Double-Blind, Sham-Controlled, Pilot Study of Trigeminal Nerve Stimulation for Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2019 Apr;58(4):403-411.e3. doi: 10.1016/j.jaac.2018.11.013. Epub 2019 Jan 28. PMID 30768393
- [Derived] Loo SK, Salgari GC, Ellis A, Cowen J, Dillon A, McGough JJ. Trigeminal Nerve Stimulation for Attention-Deficit/Hyperactivity Disorder: Cognitive and Electroencephalographic Predictors of Treatment Response. J Am Acad Child Adolesc Psychiatry. 2021 Jul;60(7):856-864.e1. doi: 10.1016/j.jaac.2020.09.021. Epub 2020 Oct 15. PMID 33068751
- See also: Pub Med Abstract — https://www.ncbi.nlm.nih.gov/pubmed/30768393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled between 04/2015 and 03/2017. Participants were recruited through community advertisements and internet postings.
Pre-assignment Details: Potential participants underwent screening and those eligible returned for baseline assessment and randomization. Of 79 individuals screened, 64 met inclusion/exclusion criteria for participation. Two of these chose not to return after screening, most likely because they were only interested in ADHD assessment.
Groups:
- Active TNS: Active TNS
  Active TNS: Participants randomized to active trigeminal nerve stimulation (TNS) administered by the Monarch eTNS System nightly during sleep.
- Sham TNS: Sham TNS
  Sham TNS: Participants randomized to sham trigeminal nerve stimulation (TNS) administered by the Monarch eTNS System nightly during sleep.
Period: 1a: 4 Week Double Blind Sham Controlled
Arm/Group | Active TNS | Sham TNS
Started | 32 | 30
Completed | 32 | 29
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: 1b: 1 Week Blinded Post Treatment
Arm/Group | Active TNS | Sham TNS
Started | 32 | 29
Completed | 31 | 28
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active eTNS: Following screening and determination of eligibility, participants at baseline are randomized to receive 4 weeks nightly treatment with active or sham eTNS, followed by one week ongoing blinded assessment following treatment discontinuation.
  Active eTNS: Participants will receive active trigeminal nerve stimulation (TNS) administered by the Monarch eTNS System nightly during sleep for 4 weeks, followed by one week of observation and followup while remaining blinded following treatment discontinuation. Participant deemed to be positive responders to blinded active treatment will be invited to continue open eTNS in a 12 month extension period.
- Sham eTNS: Following screening and determination of eligibility, participants at baseline are randomized to receive 4 weeks nightly treatment with active or sham eTNS, followed by one week ongoing blinded assessment following treatment discontinuation.
  Sham eTNS: Participants will receive sham trigeminal nerve stimulation (TNS) administered by the Monarch eTNS System nightly during sleep for 4 weeks, followed by one week of observation and followup while remaining blinded following treatment discontinuation. At the conclusion of the blinded trial, participants randomized to the sham group will be offered 4 weeks of open eTNS treatment. Participants deemed to be positive responders to open treatment will be invited to continue open nightly eTNS in a 12 month extension period.
- Total: Total of all reporting groups
Arm/Group | Active eTNS | Sham eTNS | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.26 (1.39) | 10.50 (1.37) | 10.40 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 20 | 20 | 40
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
ADHD Subtype [Count of Participants; unit: Participants] — Subtypes listed (Combined, Inattentive, Hyperactive/Impulsive) reflect different subtypes of ADHD according to diagnostic criteria. They do not reflect any grading or measure of severity.
  Participants
    Combined | 22 | 17 | 39
    Inattentive | 9 | 12 | 21
    Hyperactive/Impulsive | 1 | 1 | 2
Full Scale IQ Estimate [Mean (Standard Deviation); unit: IQ points] — Based on the Wechsler Abbreviated Scales of Intelligence, 3rd Edition.
  IQ points | 110.4 (12.3) | 107.3 (14.2) | 108.9 (13.2)
ADHD-Rating Scale Total Score [Mean (Standard Deviation); unit: units on a scale] — A dimensional rating of ADHD symptoms with scores ranging from 0 to 54, with higher scores indicating greater severity.
  units on a scale | 32.13 (6.28) | 32.83 (6.22) | 32.47 (6.21)
Clinical Global Impression - Severity [Count of Participants; unit: Participants] — A categorical measure of severity ranging from 1 ("Normal, not at all ill") to 7 ("Among the most extremely ill patients.").
  Participants
    4 (Moderately iIl) | 10 | 11 | 21
    5 (Markedly ill) | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: ADHD-IV Rating Scale (ADHD-RS)
Description: A dimensional rating of ADHD symptoms, with scores ranging from 0 - 54, and higher scores indicating greater symptom severity.
Time Frame: Change over baseline and weeks 1, 2, 3, 4 and 5.
Population: Data missing for some visits.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Active eTNS: Following screening and determination of eligibility, participants at baseline are randomized to receive 4 weeks nightly treatment with active or sham eTNS, followed by one week ongoing blinded assessment following treatment discontinuation. Positive responders will be invited to participate in a 12-month open extension.
  Active eTNS: Participants will receive active trigeminal nerve stimulation (TNS) administered by the Monarch eTNS System nightly during sleep for 4 weeks, followed by one week of observation and followup while remaining blinded following treatment discontinuation. Participant deemed to be positive responders to blinded active treatment will be invited to continue open active eTNS in a 12 month extension period.
- Sham eTNS: Following screening and determination of eligibility, participants at baseline are randomized to receive 4 weeks nightly treatment with active or sham eTNS, followed by one week ongoing blinded assessment following treatment discontinuation. Following double-blind phase, interested participants randomized to sham have an option for a 4-week open TNS trial. Positive responders will be invited to participate in a 12-month open extension.
  Sham eTNS: Participants will receive sham trigeminal nerve stimulation (TNS) administered by the Monarch eTNS System nightly during sleep for 4 weeks, followed by one week of observation and followup while remaining blinded following treatment discontinuation. At the conclusion of the blinded trial, participants randomized to the sham group will be offered 4 weeks of open eTNS treatment. Participants deemed to be positive responders to open treatment will be invited to continue open nightly active eTNS in a 12 month extension period.
Arm/Group | Active eTNS | Sham eTNS
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 32.12 (1.39) | 32.83 (1.43)
  Week 1 | 26.16 (1.39) | 28.53 (1.43)
  Week 2: number analyzed (Participants) | 32 | 29
  Week 2 | 24.74 (1.40) | 28.31 (1.48)
  Week 3: number analyzed (Participants) | 32 | 27
  Week 3 | 23.92 (1.42) | 28.78 (1.50)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 23.38 (1.40) | 27.50 (1.46)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 25.5 (1.40) | 29.1 (1.47)
Statistical Analysis 1: Comparison: Active eTNS vs Sham eTNS; Phase 1a: Outcomes were fitted via a mixed effects model with group-by-time interactions to test for treatment effects using a piecewise linear time trend. This was parameterized in the model as a standard linear variable, time (ranging from baseline to 4 weeks) and a second variable, time2, defined as 0 at baseline and time past week 1 for subsequent weeks. The time2 coefficient represents the change in slope after the initial week; Test type: Superiority; p = .54, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .38, df = 1/228
Statistical Analysis 2: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, Mixed Models Analysis — p < .05 for statistical significance; Time: F=39.97, df = 1/228
Statistical Analysis 3: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .005, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = 8.12, df = 1/228
Statistical Analysis 4: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, Mixed Models Analysis — p < .05 for statistical significance; Time2: F = 28.96, df = 1/228
Statistical Analysis 5: Comparison: Active eTNS vs Sham eTNS; Phase 1b: Outcomes were fitted via a mixed effects model with group, time, and group-by-time interactions to test for treatment effects between visits 4 and 5; Test type: Superiority; p = .02, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 6.23, df = 1/57
Statistical Analysis 6: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .05, Mixed Models Analysis — p < .05 for statistical significance; Group: F = 4.18, df = 1/57
Statistical Analysis 7: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .73, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .12, df = 1/57

2. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I)
Description: Categorical measure indicating degree improved or not improved compared with baseline for each treatment group. Minimum score = 1 (very much improved); Maximum score = 7 (very much worse). Results reflect number of participants stratified as "Improved" (CGI-I <=2) or "Not Improved" (CGI-I > 2).
Time Frame: Change over weeks 1, 2, 3, 4, and 5 compared with baseline.
Population: Data missing for some visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Active eTNS | Sham eTNS
Number analyzed (Participants) | 32 | 30
Participants
  Week 1: Improved | 8 | 4
  Week 1: Not Improved | 24 | 26
  Week 2: number analyzed (Participants) | 31 | 26
  Week 2: Improved | 12 | 4
  Week 2: Not Improved | 19 | 22
  Week 3: number analyzed (Participants) | 30 | 25
  Week 3: Improved | 14 | 3
  Week 3: Not Improved | 16 | 22
  Week 4: number analyzed (Participants) | 31 | 28
  Week 4: Improved | 16 | 4
  Week 4: Not Improved | 15 | 24
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5: Improved | 4 | 2
  Week 5: Not Improved | 27 | 26
Statistical Analysis 1: Comparison: Active eTNS vs Sham eTNS; Phase 1a: Assessed effects of group and time on categorical measure CGI-I from Baseline through Visit 4; Test type: Superiority; p = .003, Chi-squared — p < .05 for statistical significance; Group: F = 8.75, df = 1/168
Statistical Analysis 2: Comparison: Active eTNS vs Sham eTNS; Phase 1a: Assessed effects of group and time on categorical measure CGI-I from Baseline through Visit 4; Test type: Superiority; p = .17, Chi-squared — p < .05 for statistical significance; Time: F = 1.69, df = 3/168
Statistical Analysis 3: Comparison: Active eTNS vs Sham eTNS; Phase 1b: Assessed effects of group on categorical measure CGI-I from at Visit 5 compared to baseline; Test type: Superiority; p = .46, Chi-squared; Group: Chi-square = .53, df = 1

3. Secondary Outcome: Conners Global Index - Parent Report
Description: Parent completed dimensional measure of ADHD symptoms, with score range from 0- 30, and higher scores indicating more severe symptoms.
Time Frame: Change over baseline and weeks 1, 2, 3, 4, 5.
Population: Data missing for some visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active eTNS | Sham eTNS
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 18.3 (1.1) | 17.4 (1.1)
  Week 1 | 15.7 (1.1) | 16.5 (1.1)
  Week 2: number analyzed (Participants) | 32 | 29
  Week 2 | 13.0 (1.1) | 15.2 (1.2)
  Week 3: number analyzed (Participants) | 32 | 27
  Week 3 | 13.4 (1.1) | 15.2 (1.2)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 14.7 (14.7) | 14.6 (1.2)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 14.1 (1.1) | 15.7 (1.2)
Statistical Analysis 1: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .91, Mixed Models Analysis; Group: F=.01; df =1/209
Statistical Analysis 2: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .0004, Mixed Models Analysis; Time: F=13.03; df = 1/209
Statistical Analysis 3: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .37, Mixed Models Analysis; Group * time: F = .83; df = 1/209
Statistical Analysis 4: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .007, Mixed Models Analysis — Time2: F = 7.45, df = 1/209
Statistical Analysis 5: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .67, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .19, df = 1/59
Statistical Analysis 6: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .68, Mixed Models Analysis — p < .05 for statistical significance; Time: F = .17, df = 1/50
Statistical Analysis 7: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .16, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = 2.05, df = 1/50

4. Secondary Outcome: Affective Reactivity Index (ARI) - Child
Description: A child completed dimensional measure of emotional reactivity, with scores ranging from 0-12, and higher scores indicating greater severity.
Time Frame: Change over baseline and weeks 4 and 5.
Population: Data missing for some visits
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active eTNS | Sham eTNS
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 4.5 (.5) | 4.5 (.5)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 4.1 (.5) | 3.8 (.6)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 3.9 (.5) | 3.5 (.6)
Statistical Analysis 1: Comparison: Active eTNS vs Sham eTNS; Phase 1a: Outcomes were fitted via a mixed effects model with group, time, and group-by-time interactions to test for treatment effects; Test type: Superiority; p = .91, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .01, df = 1/56
Statistical Analysis 2: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .15, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 2.12, df = .15
Statistical Analysis 3: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .64, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .21, df = 1/56
Statistical Analysis 4: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .66, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .20, df = 1/59
Statistical Analysis 5: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .48, Mixed Models Analysis — p < .05 for statistical significance; Time: F = .50, df = 1/47
Statistical Analysis 6: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .81, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .06, df = 1/47

5. Secondary Outcome: Affective Reactivity Index (ARI) - Parent Report
Description: A parent completed dimensional measure of emotional reactivity, with scores ranging from 0-12, and higher scores indicating greater severity.
Time Frame: Change over baseline and weeks 4 and 5.
Population: Data missing for some visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active eTNS | Sham eTNS
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 4.4 (.6) | 4.5 (.6)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 3.6 (.6) | 3.6 (.7)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 3.8 (.7) | 4.2 (.7)
Statistical Analysis 1: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .89, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .02, df = 1/55
Statistical Analysis 2: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .14, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 2.28, df = 1/55
Statistical Analysis 3: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .80, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .06, df = .81
Statistical Analysis 4: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .93, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .01, df = 1/58
Statistical Analysis 5: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .15, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 2.22, df = 1/35
Statistical Analysis 6: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .28, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = 1.23, df = 1/35

6. Secondary Outcome: Multidimensional Anxiety Scale for Children (MASC) - Child Report
Description: A child completed rating of child anxiety, with scores ranging from 0-300, and higher scores indicating greater severity.
Time Frame: Change over baseline and weeks 4 and 5.
Population: Data missing from some visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active eTNS | Sham eTNS
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 61.0 (4.7) | 61.0 (4.9)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 59.5 (4.8) | 56.4 (4.7)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 56.1 (5.0) | 52.3 (5.3)
Statistical Analysis 1: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .91, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .01; df = 1/46
Statistical Analysis 2: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .11, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 2.62, df = 1/46
Statistical Analysis 3: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .40, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .71; df = .40
Statistical Analysis 4: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .49, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .48. df = 1/55
Statistical Analysis 5: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .18, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 1.87, df = 1/55
Statistical Analysis 6: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .72, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .13, df = 1/38

7. Secondary Outcome: Multidimensional Anxiety Scale for Children (MASC) - Parent Report
Description: A parent completed rating of child anxiety, with scores ranging from 0-300, and higher scores indicating greater severity.
Time Frame: Change over baseline and weeks 4 and 5.
Population: Data missing for some visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active eTNS | Sham eTNS
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 46.2 (3.0) | 48.4 (3.1)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 33.9 (3.0) | 42.9 (3.2)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 32.4 (2.9) | 38.2 (3.0)
Statistical Analysis 1: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .62, Mixed Models Analysis; Group: F =.25, df = 1/53
Statistical Analysis 2: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .06, Mixed Models Analysis; Time: F = 3.58, df = 1/53
Statistical Analysis 3: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .09, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = 2.90, df 1/53
Statistical Analysis 4: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .06, Mixed Models Analysis — p < .05 for statistical significance; Group: F = 3.36, df = 1/58
Statistical Analysis 5: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .05, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 4.20, df = 1/31
Statistical Analysis 6: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .42, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .66, df = 1/31

8. Secondary Outcome: Height
Description: A dimensional measure assessed in centimeters (cm).
Time Frame: Change over baseline and weeks 1, 4, and 5.
Population: Data missing for some visits.
Measure: Least Squares Mean (Standard Error); unit: cm.
Arm/Group | Active TNS | Sham TNS
Number analyzed (Participants) | 32 | 30
cm.
  Baseline | 142.82 (1.78) | 141.45 (1.84)
  Week 1 | 142.79 (1.78) | 141.57 (1.84)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 143.14 (1.78) | 142.31 (1.84)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 143.58 (1.81) | 142.30 (1.90)
Statistical Analysis 1: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .29, Mixed Models Analysis — p < .05 for statistical significance; Group: F = 0.29, df = 1/129
Statistical Analysis 2: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .02, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 5.83, df = 1/129
Statistical Analysis 3: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .31, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = 1.03, df = 1/129
Statistical Analysis 4: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .69, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .16, df = 1/59
Statistical Analysis 5: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .33, Mixed Models Analysis — p < .05 for statistical significance; Time: F = .98, df = 1/54
Statistical Analysis 6: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .35, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .88, df = 1/54

9. Secondary Outcome: Weight
Description: A dimensional measure assessed in kilograms (kg).
Time Frame: Change over baseline and weeks 1, 4, and 5.
Population: Data missing for some visits.
Measure: Least Squares Mean (Standard Error); unit: kg.
Arm/Group | Active eTNS | Sham eTNS
Number analyzed (Participants) | 32 | 30
kg.
  Baseline | 38.83 (1.88) | 35.34 (1.95)
  Week 1 | 39.12 (1.88) | 35.58 (1.95)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 39.65 (1.88) | 35.67 (1.95)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 39.85 (1.93) | 35.71 (2.03)
Statistical Analysis 1: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .21, Mixed Models Analysis — p < .05 for statistical significance; Group: F = 1.62, df = 1/128
Statistical Analysis 2: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .02, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 5.18, df = 1/128
Statistical Analysis 3: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .01, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = 6.89, df = 1/128
Statistical Analysis 4: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .15, Mixed Models Analysis — p < .05 for statistical significance; Group: F= 2.16, df = 1/59
Statistical Analysis 5: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .05, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 4.15, df = 1/55
Statistical Analysis 6: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .79, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .07, df = 1/55

10. Secondary Outcome: Systolic Blood Pressure
Description: A dimensional measure expressed in mm mercury (Hg).
Time Frame: Change over baseline and weeks 1, 4, and 5.
Population: Data missing from some visits.
Measure: Least Squares Mean (Standard Error); unit: mm Hg.
Arm/Group | Active TNS | Sham TNS
Number analyzed (Participants) | 32 | 30
mm Hg.
  Baseline | 108.50 (2.26) | 106.10 (2.36)
  Week 1 | 107.03 (2.26) | 109.20 (2.34)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 111.00 (2.26) | 107.79 (2.36)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 112.26 (2.02) | 106.10 (2.13)
Statistical Analysis 1: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .94, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .01, df = 1/128
Statistical Analysis 2: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .76, Mixed Models Analysis — p < .05 for statistical significance; Time: F = .09, df = 1/128
Statistical Analysis 3: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .39, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .75, df =1/128
Statistical Analysis 4: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .09, Mixed Models Analysis — p < .05 for statistical significance; Group: F = 3.06, df = 1/59
Statistical Analysis 5: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .79, Mixed Models Analysis — p < .05 for statistical significance; Time: F = .07, df = 1/55
Statistical Analysis 6: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .22, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = 1.55, df = 1/55

11. Secondary Outcome: Diastolic Blood Pressure
Description: A dimensional measure assessed in mm mercury (Hg).
Time Frame: Change over baseline and weeks 1, 4, and 5.
Population: Data missing for some visits.
Measure: Least Squares Mean (Standard Error); unit: mm Hg.
Arm/Group | Active TNS | Sham TNS
Number analyzed (Participants) | 32 | 30
mm Hg.
  Baseline | 64.97 (1.66) | 63.61 (1.73)
  Week 1 | 63.69 (1.66) | 62.33 (1.71)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 65.09 (1.66) | 61.01 (1.73)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 65.30 (1.76) | 60.89 (1.86)
Statistical Analysis 1: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .64, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .22, df = 1/128
Statistical Analysis 2: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .19, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 1.49, df = 1/128
Statistical Analysis 3: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .22, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = 1.49, df = 1/128
Statistical Analysis 4: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .05, Mixed Models Analysis — p < .05 for statistical significance; Group: F = 3.95, df = 1/59
Statistical Analysis 5: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .96, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 0.00, df = 1/55
Statistical Analysis 6: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .92, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = .01, df = 1/55

12. Secondary Outcome: Pulse
Description: Heart rate in beats per minute (bpm).
Time Frame: Change over baseline and weeks weeks 1, 4, and 5.
Population: Data missing for some visits.
Measure: Least Squares Mean (Standard Error); unit: bpm.
Arm/Group | Active TNS | Sham TNS
Number analyzed (Participants) | 32 | 30
bpm.
  Baseline | 76.69 (2.27) | 76.70 (2.37)
  Week 1 | 79.91 (2.27) | 79.70 (2.34)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 81.78 (2.27) | 75.18 (2.37)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 79.42 (2.10) | 78.18 (2.22)
Statistical Analysis 1: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .79, Mixed Models Analysis — p < .05 for statistical significance; Group: F = .07, df = 1/128
Statistical Analysis 2: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .30, Mixed Models Analysis — p < .05 for statistical significance; Time: F = 1.10, df = 1/128
Statistical Analysis 3: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .03, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = 4.61, df = 1/128
Statistical Analysis 4: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .14, Mixed Models Analysis — p < .05 for statistical significance; Group: F = 2.24, df = 1/59
Statistical Analysis 5: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .82, Mixed Models Analysis — p < .05 for statistical significance; Time: F = .05, df = 1/55
Statistical Analysis 6: Comparison: Active TNS vs Sham TNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .07, Mixed Models Analysis — p < .05 for statistical significance; Group * time: F = 3.35, df = 1/55

13. Secondary Outcome: Children's Depression Inventory (CDI)
Description: A child completed self-report dimensional measure of depressive symptoms, with range of scores from 0 to 54. Higher scores reflect increasing depression. Cutoff scores < 17 to 20 are generally considered to be in the normative range. A score of 36 or higher reflects a relatively severe depression.
Time Frame: Change over baseline and weeks 4 and 5.
Population: Data missing for some visits.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active eTNS | Sham eTNS
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 10.14 (1.23) | 9.10 (1.23)
  Week 4: number analyzed (Participants) | 32 | 29
  Week 4 | 8.94 (1.22) | 8.21 (1.24)
  Week 5: number analyzed (Participants) | 31 | 28
  Week 5 | 7.88 (1.32) | 7.34 (1.37)
Statistical Analysis 1: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = .55, Mixed Models Analysis; Group: F = .36, df = 1/52
Statistical Analysis 2: Comparison: Active eTNS vs Sham eTNS; Phase 1a: Outcomes were fitted via a mixed model with group, time, and group-by-time interactions to test for treatment effects; Test type: Superiority; p = .34, Mixed Models Analysis; Time: F = .09, df = 1/52
Statistical Analysis 3: Comparison: Active eTNS vs Sham eTNS; Phase 1 a: Outcomes were fitted via a mixed effects model with group, time, and group-by-time interaction to test for treatment effects; Test type: Superiority; p = .81, Mixed Models Analysis; Group * time: F = .06, df = 1/52
Statistical Analysis 4: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .83, Mixed Models Analysis; Group: F = .05, df = 1/59
Statistical Analysis 5: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .04, Mixed Models Analysis; Time: F = 4.52, df = 1/43
Statistical Analysis 6: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .73, Mixed Models Analysis; Group * time: F = .12, df = 1/43

14. Secondary Outcome: Conners Global Index - Teacher
Description: Teacher completed dimensional measure of ADHD symptoms, with scores ranging from 0-30, and higher scores indicating more severe symptoms.
Time Frame: Change over baseline and weeks 1, 2, 3, 4, 5.
Population: Results may not be valid due to problems with data collection leading to substantial missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active eTNS | Sham eTNS
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline: number analyzed (Participants) | 13 | 11
  Baseline | 15.76 (1.32) | 15.15 (1.32)
  Week 1: number analyzed (Participants) | 17 | 11
  Week 1 | 15.86 (1.23) | 11.37 (1.46)
  Week 2: number analyzed (Participants) | 15 | 6
  Week 2 | 14.36 (1.27) | 15.64 (1.77)
  Week 3: number analyzed (Participants) | 9 | 5
  Week 3 | 14.56 (1.92) | 16.56 (1.92)
  Week 4: number analyzed (Participants) | 6 | 5
  Week 4 | 15.43 (1.69) | 14.53 (1.89)
  Week 5: number analyzed (Participants) | 3 | 2
  Week 5 | 11.54 (3.33) | 18.83 (3.89)
Statistical Analysis 1: Comparison: Active eTNS vs Sham eTNS; Phase 1a: Outcomes were fitted via a mixed effects model with group-by-time interactions to test for treatment effects using a piecewise linear time trend. This was parametrized in the model as a standard linear viable, time (ranging from baseline to 4 weeks) and a second variable, time2. defined as 0 at baseline and time past week 1 for subsequent weeks. The time 2 coefficient represents the change in slope after the initial week; Test type: Superiority; p = .21, Mixed Models Analysis; Group: F = 1.62, df = 1/58
Statistical Analysis 2: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = .39, Mixed Models Analysis; Time: F = .74, df = 1/58
Statistical Analysis 3: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = .18, Mixed Models Analysis; Time2: F = 1.88, df = 1/58
Statistical Analysis 4: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = .22, Mixed Models Analysis; Group * time: F = 1.56; df = 1/58
Statistical Analysis 5: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = .21, Mixed Models Analysis; Group: F = 1.72, df = 1/12
Statistical Analysis 6: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 1, Mixed Models Analysis — Test not valid due to insufficient data; Time: F = 0.00, df = 1/0
Statistical Analysis 7: Comparison: Active eTNS vs Sham eTNS; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 1, Mixed Models Analysis — Test not valid due to insufficient data; Group * time: F = .87, df = 1/0

15. Other Pre Specified Outcome: Affective Posner Task
Description: A laboratory measure of frustration tolerance.
Time Frame: Baseline, and Weeks 1 and 4
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Attention Network Task (ANT) Response Inhibition
Description: A computer-administered laboratory measure of executive function.
Time Frame: Baseline, Weeks 1 and 4
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Spatial Working Memory (SWM)
Description: A computer-administered laboratory measure of executive function.
Time Frame: Baseline, Weeks 1 and 4
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Electroencephalography (EEG)
Description: A laboratory measure of cortical activity.
Time Frame: Baseline and Week 4
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Behavior Rating Inventory of Executive Functioning (BRIEF)
Description: A parent completed rating of child executive function. Comprises 5 sub scales that measure various measures of behavior and cognition. Raw scores on each measure are converted to T scores ranging from 28 to 103, with higher scores indicating greater difficulties.
Time Frame: Baseline, end of Weeks 4 and 5.
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Children's Sleep Habits Questionnaire (CSHQ)
Description: A parent completed 33-item scale to assess sleep related problems. Total scores range from 33 to 99 divided among 8 sub scales , with higher scores indicating more severe difficulties.
Time Frame: Weekly for double-blind trial.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data were collected over the double-blind study, beginning at baseline and then weekly for 5 weeks.
Description: Adverse events were solicited via a structured side effects questionnaire and open inquiry completed at baseline and each weekly visit during the double-blind phases.
Arm/Group | Active TNS | Sham TNS
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 23/32 | 22/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TNS (N=32) | Sham TNS (N=30)
Trouble sleeping (Psychiatric disorders) | 6 (11) | 5 (6)
Nightmares (Psychiatric disorders) | 2 (2) | 0 (0)
Drowsy (Nervous system disorders) | 7 (9) | 4 (5)
Hyperactive (Psychiatric disorders) | 13 (27) | 19 (40)
Feels strange (Psychiatric disorders) | 0 (0) | 2 (2)
Tingling (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (7)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (2)
Slurred speech (Nervous system disorders) | 0 (0) | 1 (1)
Rapid heartbeat (Cardiac disorders) | 1 (1) | 0 (0)
Trouble catching breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomachache (Gastrointestinal disorders) | 2 (2) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (6) | 3 (10)
Frequent urination (Renal and urinary disorders) | 2 (5) | 0 (0)
Frequent sweating (Nervous system disorders) | 1 (1) | 1 (1)
Decreased appetite (General disorders) | 1 (1) | 1 (1)
Increased appetite (General disorders) | 6 (13) | 2 (2)
Difficulty finding words (Nervous system disorders) | 0 (0) | 3 (6)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Apathy (Psychiatric disorders) | 2 (2) | 3 (3)
Clenching teeth (Psychiatric disorders) | 4 (6) | 3 (3)
Fatigue (General disorders) | 4 (4) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Wish to be dead. (Psychiatric disorders) | 0 (0) | 0 (0) — Based on Columbia-Suicide Severity Rating Scale (C-SSRS)
Non-specific active suicidal thoughts (Psychiatric disorders) | 0 (0) | 0 (0) — Based on Columbia-Suicide Severity Rating Scale (C-SSRS)
Active suicidal ideation without intent (Psychiatric disorders) | 0 (0) | 0 (0)
Active suicidal ideation with some intent (Psychiatric disorders) | 0 (0) | 0 (0) — Based on Columbia-Suicide Severity Rating Scale (C-SSRS)
Active suicidal ideation with active plan and intent (Psychiatric disorders) | 0 (0) | 0 (0) — Based on Columbia-Suicide Severity Rating Scale (C-SSRS)

LIMITATIONS AND CAVEATS:
Insufficient data were collected with the Conners Teacher Report leading to small number of participants analyzed. Results are likely not valid.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT02155608/Prot_SAP_000.pdf
  • Informed Consent Form (2015-04-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT02155608/ICF_001.pdf